CLINICAL TRIAL: NCT05335486
Title: Investigating RELEARN Neurofeedback as Treatment for Chronic Musculoskeletal Pain
Acronym: RELEARN
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of clinician interest and insufficient patient availability
Sponsor: Redo-Neurosystems (Industry)
Collaborators: Regionshospital Nordjylland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELEARN2200701
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Chronic Knee Pain; Chronic Pain; Osteoarthritis
Keywords: chronic pain; Chronic Knee Pain; Osteoarthritis; Neurofeedback; EEG; EMG; Movement evoked potentials; Neuroplasticity; Pain perception
MeSH Terms: conditions — Chronic Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELEARN - Intervention (Experimental): Intervention group participants will be seen at the orthopedic ward and receive standard care for knee osteoarthrosis, defined by Danish clinical guidelines.
  In addition, intervention group participants will be asked to attend eight sessions of RELEARN neurofeedback with an approximate duration of 45 minutes per session. Also, participants will undergo three follow-up sessions: one month, three months, and five months post-intervention
  Interventions: Device: RELEARN Neurofeedback
- Standard care control (Active Comparator): Standard Care control. Control group participants will be seen at the orthopedic ward and receive standard care for knee osteoarthrosis, defined by Danish clinical guidelines. During standard care, the control group participants will be asked to attend eight control sessions with no RELEARN intervention with an approximate duration of 5 minutes per session. Also, participants will undergo three follow-up sessions: one month, three months, and five months post-intervention
  Interventions: Other: Standard care control

INTERVENTIONS:
Device: RELEARN Neurofeedback — Standard care + The RELEARN intervention.
  Intervention group participants will be seen at the orthopedic ward and receive standard care for knee osteoarthrosis, defined by Danish clinical guidelines.
  During standard care, intervention group participants will be subject to the RELEARN intervention, consisting of encephalography (EEG) neurofeedback of cerebral movement evoked signatures of pain, where the participants will be instructed in attempting to manipulate these signatures to reduce pain perception.
  Arms: RELEARN - Intervention
Other: Standard care control — Standard Care control.
  Control group participants will be seen at the orthopedic ward and receive standard care for knee osteoarthrosis, defined by Danish clinical guidelines. During standard care, the control group participants will be asked to attend eight control sessions with no RELEARN intervention with an approximate duration of 5 minutes per session. Also, participants will undergo three follow-up sessions: one month, three months, and five months post-intervention
  Arms: Standard care control

SUMMARY:
This clinical investigation will be carried out as a randomized controlled trial conducted at the Northern Regional Hospital, Hjørring. This investigation will enrol 36 patients suffering from severe knee osteoarthritis pain, primarily from the orthopaedic ward at Hjørring Hospital, where potential participants will be identified during routine consultations.

The RELEARN intervention consists of encephalography (EEG) neurofeedback of cerebral movement evoked signatures of pain, where the participants will be instructed in attempting to manipulate these signatures to reduce pain perception. This investigation is carried out to analyse the clinical performance and safety of the RELEARN neurofeedback software.

DETAILED DESCRIPTION:
The participants will be randomized into treatment group A and control group B, 1:1 and be stratified based on age, sex, and ethnicity. Group A participants will be asked to attend eight sessions of RELEARN neurofeedback with an approximate duration of 45 minutes per session, and group B participants will be asked to attend eight sessions with no intervention and serve as no-treatment controls with an approximate duration of 5 minutes per session. Both groups (A and B) will undergo three follow-up sessions: one month, three months, and five months post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Knee arthrosis (Kellgren-Lawrence score of ≥ 2)
3. 24h VAS ≥ 4
4. Ongoing pain, lasting more than three months

   Exclusion Criteria:

   Participants who meet any of the below criteria will be excluded from the investigation:
5. Pregnant or lactating woman
6. Use of opioids or cannabis
7. Active drug addiction defined as the use of cannabis, opioids, or other drugs
8. Previous or current neurologic, systemic, or mental illness, including any liver, kidney or metabolic disease.
9. Rheumatoid arthritis
10. Evidence of other pain types such as visceral, neuropathic, or malignant pain.
11. Evidence of other sources of ongoing pain such as root affect, traumas, or congenital malformation
12. Severe inflammation in the area of interest
13. Blindness or deafness
14. Consumption of alcohol, caffeine, nicotine on test day
15. Recent history of fractures or surgery in the area of interest
16. Participation in other clinical trials throughout the study period and one month prior to participation
17. History of epilepsy
18. Obesity class III and above. I.e. BMI > 39,9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Perception | Up to 6 month
  Change in the 10-point Visual Analogue Scale (VAS) over time (0 = no pain, 10 = maximum imaginable pain)

SECONDARY OUTCOMES:
Change in quality of life | Up to 6 month
  QoL (EQ-5D), Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Change in pain characteristics | Up to 6 month
  Pain characteristics (MPQ and WOMAC)
Change in consumption of analgesics | Up to 6 month
  Consumption of analgesics (MQS-III)
Evaluate the safety of the RELEARN software by assessment of adverse events and device deficiencies | Up to 6 month
  Incidence of AE/ADE/SAE/SADE/DD

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christian Leutscher, Dr. PhD, Principal Investigator — Center of Clinical Research, Regional Hospital North Jutland, Hjørring, Denmark
Locations (1):
- Center for Clinical Research, Hjørring, Denmark

IPD SHARING:
Plan to Share IPD: No